CLINICAL TRIAL: NCT03762226
Title: Influence of Systemic Parameters in Diabetic Macular Edema - LIPSIA Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, PD Dr. habil. Matus Rehak, Prof. MUDr. Matus Rehak, University of Leipzig
Other Study IDs: 72311607
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Diabetic Macular Edema; Macular Edema; Retinal Vein Occlusion
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Serum and heparine blood sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with Macular edema: Patients with clinically significant macular edema due to diabetes or retinal vein occlusion, undergoing at least 4 monthly intravitreal anti-VEGF injections.
  Interventions: Drug: Anti-VEGF

INTERVENTIONS:
Drug: Anti-VEGF — Patients will undergo as part of the routine care 4 monthly anti-VEGF injections.
  Other Names: Intravitreal anti-VEGF injection

SUMMARY:
This study aims to evaluate the influence and prognostic value of systemic factors (such as the cardiovascular and metabolic status) on the treatment response to anti-VEGF therapy in macular edema due to diabetes or retinal vein occlusion.

DETAILED DESCRIPTION:
This study includes patients with macular edema (ME) due to diabetes or retinal vein occlusion in the need of treatment.

At baseline patients underwent an extensive ophthalmological examination (best-corrected visual acuity, OCT, OCT-angiography, fluorescein angiography, fundus photography). Besides that, systemic work-up (including 24h blood pressure measurement, electrocardiogram, and serological blood testing) is conducted.

Patients underwent routine ME treatment including at least 4 monthly anti-VEGF injections, as first-line therapy. Further injections will be conducted if needed. Re-treatment criteria are: persistent intra- and/or subretinal fluid seen on SD-OCT, central subfield thickness > 300 µm. Ophthalmological examination will be repeated at month 3, 6 and month 12. Systemic work-up will be repeated at month 6.

Primary outcome is the correlation of systemic parameters with functional and anatomical response at month 6. Secondary outcome is the correlation of systemic parameters with functional and anatomical response at month 12.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years
2. Diagnosis of diabetes mellitus (type 1 or type 2) and/or retinal vein occlusion
3. macular edema causing visual loss, with study eye VA of 0.1 - 1.0 logMAR (20/25 - 20/200 Snellen equivalent)
4. macular edema defined clinically and by retinal thickness of > 300 µm in the central subfield thickness (CST) with intra +/- subretinal fluid seen on spectral domain optical coherence tomography
5. last intravitreal treatment > 3 months ago.

Exclusion Criteria:

1. concomitant ocular disease that could cause macular edema (including choroidal neovascularization from any cause, uveitis or intraocular surgery less than 6 months ago).
2. any concomitant ocular or neurological condition that could affect Vision except of cataract.
3. pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with macular edema due to Diabetes or retinal vein occlusion
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of systemic factors on functional and anatomical outcome at month 6. | 6 months
  Correlation between blood pressure and serological Parameters at baseline and visual acuity/central subfield thickness at month 6.

SECONDARY OUTCOMES:
Correlation of systemic factors on functional and anatomical outcome at month 12. | 12 months
  Correlation between blood pressure and serological parameters at baseline and visual acuity/central subfield thickness at month 12.

CONTACTS AND LOCATIONS:
Overall Officials: Matus Rehak, MD, PhD, Principal Investigator — University Hospital Leipzig, Department of Ophthalmology
Locations (1):
- University Hospital Leipzig, department of ophthalmology, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No